CLINICAL TRIAL: NCT06599385
Title: Platelet Transfusion in Critically Ill Patients With Thrombocytopenia
Acronym: TRAMPOLINE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APHP230835
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Thrombocythemia
Keywords: Platelet transfusion; Thrombocythemia
MeSH Terms: conditions — Thrombocytosis

STUDY DESIGN:
Intervention Model Description: Prospective non-inferiority open-label randomised trial with two comparative groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-threshold (Active Comparator)
  Interventions: Other: Platelet transfusion if platelet count ≤ 10 G/L
- High threshold (Experimental)
  Interventions: Other: Platelet transfusion when platelet count ≤ 20 G/L

INTERVENTIONS:
Other: Platelet transfusion if platelet count ≤ 10 G/L — Platelet transfusion as soon as platelet count falls ≤ 10 G/L
  Arms: Low-threshold
Other: Platelet transfusion when platelet count ≤ 20 G/L — Platelet transfusion will be initiated immediately after randomisation
  Arms: High threshold

SUMMARY:
Thrombocytopenia is a common biological disorder in critically ill patients. The main supportive treatment is platelet transfusion with the aim of preventing and treating bleeding and securing invasive procedures. Current guidelines suggest that prophylactic platelet transfusion should probably be administered in non-bleeding critically ill patients at platelet count triggers of 10 to 20 G/L, albeit with very low certainty since extrapolated from studies carried out in stable patients with hematological malignancies. Indications for prophylactic platelet transfusion have not been properly addressed in adult ICU patients with regard to their particular risk of bleeding and prognosis. We propose the TRAMPOLINE study in order to address two different platelet count thresholds of 10 G/L (low threshold) or 20 G/L (high threshold) for the prevention of ICU-acquired bleeding in critically ill patients with severe thrombocytopenia.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 y.o. AND
2. Hospitalisation in the ICU with at least one of the following life support during the current ICU stay (past or ongoing, regardless of indications)

   * circulatory support (inotropes/ vasopressors at any dose)
   * respiratory support (invasive mechanical ventilation, non-invasive ventilation, continuous positive airway pressure (CPAP), high-flow nasal oxygen, O2 supply ≥ 6 L/min)
   * renal replacement therapy for metabolic disturbances and/or acute and acute-on chronic kidney failure (if not previously under chronic hemodialysis) AND
3. Platelet count ≤ 20 G/L within the last 24h (first occurrence at any time during the ICU stay) AND
4. expected ICU stay for at least 48 hours from the time of enrollment AND
5. Signed consent by the patient or his/her relative, or under an emergency procedure (emergency enrollment notified in the medical file, with requirement for confirmation consent a posteriori)

Exclusion Criteria:

1. Major bleeding (WHO grade 3-4) or mild bleeding (WHO grade 2) within the present hospitalization
2. Major surgery within the recent 72 hours
3. Intracranial or retinal bleeding within the recent 7 days
4. Non- or contra-indication to prophylactic platelet transfusion (immune thrombocytopenia, thrombotic microangiopathy)
5. Indications for increased prophylactic platelet transfusion threshold > 20 G/L (conditions associated with increased risk of bleeding including, but not limited to extra-corporeal membrane oxygenation, therapeutic anticoagulant treatment, fibrinolysis…)
6. Known full refractory status to platelet transfusion (prophylactic transfusion not recommended)
7. Prophylactic platelet transfusion already applied at platelet count ≤ 20 G/L during the present ICU stay
8. Patient opposed to transfusion of blood products
9. Moribund patients (death expected within the next 24 hours)
10. Pregnancy/breastfeeding
11. Not covered by French Social Security (health insurance)
12. Patient under safeguarding of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 536 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of ICU-acquired severe and debilitating bleeding | Until ICU discharge or up to 28 days in ICU
  Grades 3-4 of the modified WHO bleeding scale, assessed during the ICU stay, from the time of randomization to ICU discharge (or to the end of 28-day intervention period in patients remaining in the ICU after 28 days). Bleeding events will be collected up to 72h after ICU discharge.
  The modified WHO bleeding scale, commonly used in observational studies and trials to assess the severity of bleeding. It comprises 4 grades: grade 1 (minor blood loss), grade 2 (mild blood loss), grade 3 (severe blood loss (most often requiring Red Blood Cell transfusion) and grade 4 (debilitating blood loss).

SECONDARY OUTCOMES:
Incidence of ICU-acquired mild bleeding | Until ICU discharge or at 28 days in ICU
  WHO grade 2
Incidence of ICU-acquired mild to debilitating bleeding | Until ICU discharge or up to 28 days in ICU
  WHO grade 2-3-4
Total number of platelet transfusions episodes | Until ICU discharge or up to 28 days in ICU
Number of prophylactic platelet transfusions episodes | Until ICU discharge or up to 28 days in ICU
Doses of transfused platelets | Until ICU discharge or up to 28 days in ICU
Number of packed red cell transfusions | Until ICU discharge or up to 28 days in ICU
Volumes of packed red cell transfusions | Until ICU discharge or up to 28 days in ICU
Volumes of fresh frozen plasma | Until ICU discharge or up to 28 days in ICU
Incidence of ICU-acquired infections | Up to 72 hours after ICU discharge
Incidence of acquired arterial thrombotic events | Up to 72 hours after ICU discharge
  Acute coronary syndrome, acute limb ischemia, mesenteric ischemia, stroke
Incidence of acquired venous thrombotic events | Up to 72 hours after ICU discharge
  Thrombophlebitis and pulmonary embolism
Incidence of Central Venous Catheter (CVC)-related hemorrhagic and infectious complications | Up to 72 hours after ICU discharge
Incidence of platelet transfusion-related side effects | Up to 72 hours after ICU discharge
  Any significant transfusion reaction such as chills and fever or side effect requiring to be reported to the local hemovigilance system
Incidence of transfusion-related pulmonary manifestations (acute pulmonary oedema and acute lung injury (TRALI)) | Up to 72 hours after ICU discharge
Incidence of anti-HLA/HPA immunization | Up to 72 hours after ICU discharge
  Investigated in case of platelet transfusion refractoriness
In ICU survival | Up to 90 days
  Investigated in case of platelet transfusion refractoriness
In hospital survival | Up to 90 days
  Investigated in case of platelet transfusion refractoriness
28 day survival | At 28 days
  Investigated in case of platelet transfusion refractoriness
In ICU length of stay | Up to 90 days
In hospital length of stay | Up to 90 days
90-day survival | Up to 90 days
90-day hospital costs | Up to 90 days
  From randomization to day 90

IPD SHARING:
Plan to Share IPD: Undecided